CLINICAL TRIAL: NCT02303912
Title: Phase 1B Open Label Study to Assess the Safety, Pharmacokinetics and Clinical Activity of Nuc-1031 Given on Days 1 & 8 With Carboplatin on Day 1, q3-weekly for 6 Cycles in Participants With Recurrent Ovarian Cancer.
Brief Title: Safety and Efficacy Study of Nuc-1031 and Carboplatin Combination to Treat Recurrent Ovarian Cancer
Acronym: ProGem2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-002; 2014-002006-21 (EudraCT Number)
Record Dates: First submitted 2014-10-10; First posted 2014-12-01 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Recurrent Ovarian Cancer
Keywords: relapsed epithelial ovarian cancer,; relapsed fallopian tube cancer; relapsed primary peritoneal cancer.
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — NUC-1031; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label dose escalation (Other): Nuc-1031 IV injection on day 1 and day 8 repeated every 21 days Carboplatin IV infusion on day 1 repeated every 21 days.
  Dose escalation will be done using 3+3 dose escalation design
  Interventions: Drug: Nuc-1031 and Carboplatin

INTERVENTIONS:
Drug: Nuc-1031 and Carboplatin — Nuc-1031 IV injection on day 1 and day 8 repeated every 21 days Carboplatin IV infusion on day 1 repeated every 21 days (Total 6 cycles)

SUMMARY:
A first in human experimental treatment in which an experimental medicine,Nuc-1031, is used in combination with a standard cancer medicine, carboplatin, to treat ovarian cancer which reappear after standard cancer treatment. The aim of the trial is to determine safety, effectiveness, and clinical activity of this combination treatment.

DETAILED DESCRIPTION:
Nuc-1031 and carboplatin combination is a new experimental treatment for ovarian cancer which reappear after standard chemotherapy. Chemotherapy is the name for drug treatments to kill or control the growth of cancer cells. Although there is some evidence from laboratory and clinical studies that Nuc-1031 is effective in the treatment of ovarian cancer, it has not yet been tested in combination with another chemotherapy drug. So this combination treatment is classed as a first in human study(Phase1B). The aim of the study is to investigate whether adding Nuc-1031 to carboplatin can improve the benefits of chemotherapy.

Other purposes are to find out whether Nuc-1031 is safe to give with carboplatin, to identify the correct dose of Nuc-1031 when given with carboplatin and establish how effective the combination is at treating ovarian cancer. This study is also designed to enable us to find out whether Nuc-1031 adds further benefit, over and above that achieved by carboplatin alone, when treating ovarian cancer. and carboplatin combination will be given in six cycles. Each cycle is 3 weeks long. On first day of first week of each cycle (day1), selected study participants will receive one dose of both Nuc-1031 and Carboplatin chemotherapy. Following this, the study participant will receive a second dose of Nuc-1031 alone on first day of second week (day 8). This schedule will be repeated every 3 weeks for 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed written informed consent.
* Original diagnosis and/or histological confirmation of relapsed epithelial ovarian, fallopian tube or primary peritoneal cancer.
* Relapse ≤24 months from completion of platinum (carboplatin or cisplatin) or platinum-containing regimen.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Measurable disease as defined by Response Evaluation Criteria In Solid Tumours (RECIST) criteria version 1.1; January 2009 and/or evaluable disease (evaluable: cytologically or radiologically detectable disease such as ascites, peritoneal deposits, or lesions which do not fulfill RECIST criteria version 1.1 for measurable disease) [1,2]. Participants for whom disease and response to therapy can be monitored by serum Cancer Antigen 125 (CA125) levels will also be eligible.
* Adequate bone marrow function as defined by: White Blood Cells of ≥ 3 x109/L, Absolute Neutrophil Count (ANC) of ≥ 2.0 x 109/L, platelet count of ≥ 100.0 x 109/L, and haemoglobin of ≥ 9 g/dL.
* Adequate liver function, as determined by: Serum total bilirubin ≤1.5 x Upper Limit of Normal [(ULN), Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 2.5 x ULN, albumin ≥ 30g/L.
* Adequate renal function assessed as glomerular filtration rate(GFR) ≥ 60 mL/min using Cr51-ethylenediaminetetraacetic acid (EDTA) method.
* Ability to comply with protocol requirements.
* Participants must be postmenopausal (12 months of amenorrhea), surgically sterile or they must agree to use a physical method of contraception. Oral or injectable contraceptive agents cannot be the sole method of contraception. Participants of child-bearing potential must have a negative serum pregnancy test within seven days prior to the first study drug administration.

Exclusion Criteria:

* History of allergic reactions attributed to previous gemcitabine treatment.
* Previous treatment with Nuc-1031.
* History of allergic reactions attributed to previous carboplatin treatment.
* Symptomatic Central Nervous System (CNS) or leptomeningeal metastases.
* Prior chemotherapy, radiotherapy (other than short cycle of palliative radiotherapy for bone pain), or immunotherapy within 28 days of first receipt of study drug (within 6 weeks for nitrosoureas and mitomycin C). Hormone therapy within 14 days of first receipt of study drug.
* Prior toxicities from chemotherapy or radiotherapy which have not regressed to Grade ≤ 1 severity [National Cancer Institute -Common Terminology Criteria for Adverse Events, (NCI-CTCAE) version 4.03] except for neuropathy and alopecia.
* Another active cancer (excluding basal cell carcinoma) within the last 3 years.
* Participants with uncontrolled concomitant illness or active infection requiring IV antibiotics.
* Participants with serious illnesses, medical conditions, or other medical history, including laboratory results, which, in the investigator's opinion, would be likely to interfere with a their participation in the study, or with the interpretation of the results.
* Known Human Immunodeficiency Virus (HIV) or known active Hepatitis B or C.
* Any condition (e.g., known or suspected poor compliance, psychological instability, geographical location, etc.) that, in the judgment of the investigator, may affect the participant's ability to sign the informed consent and undergo study procedures.
* Currently pregnant, lactating or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-11; Primary Completion 2017-01-23 (Actual); Study Completion 2017-01-23 (Actual)

PRIMARY OUTCOMES:
To determine the Recommended Phase II Dose (RP2D) of Nuc-1031 and carboplatin when administered in combination. | 1 year

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of Nuc-1031 administered in combination with carboplatin measured by adverse events (AE) and changes from baseline in vital signs, clinical laboratory parameters, and electrocardiography (ECG) assessments. | 1 year
To evaluate the objective response rate (ORR) of Nuc-1031 administered in combination with carboplatin in participants with recurrent ovarian cancer. | 1 year
To evaluate the clinical benefit rate (CBR) of Nuc-1031 administered in combination with carboplatin in participants with recurrent ovarian cancer. | 1 year
To evaluate the progression free survival (PFS) of participants with recurrent ovarian cancer treated with Nuc-1031 in combination with carboplatin. | 1 year
To evaluate Overall Best Response, utilising the evaluation criteria determined by the Gynecologic Cancer Intergroup (GCIG), combining the change in CA125 from baseline with RECIST 1.1 assessment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Blagden, MBBS, MRCP, Study Director — University of Oxford
Locations (1):
- Garry Weston Cancer Centre, Hammersmith Hospital, London, United Kingdom